CLINICAL TRIAL: NCT04571034
Title: Effects of Roller Massage on Short-Term Passive Muscle Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey Sykora (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Sykora, Study Coordinator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 60480
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Muscle Tightness
Keywords: massage; roller; quadriceps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Sham Comparator): Healthy adults receiving sham comparator.
  Interventions: Procedure: Sham Therapeutic Ultrasound
- Medium-Intensity Roller Massage (Experimental): Healthy adults receiving medium-intensity roller massage.
  Interventions: Procedure: Medium-Intensity Roller Massage
- High-Intensity Roller Massage (Experimental): Healthy adults receiving high-intensity roller massage.
  Interventions: Procedure: High-Intensity Roller Massage

INTERVENTIONS:
Procedure: Sham Therapeutic Ultrasound — A standard ultrasound machine (Vectratm by Chattanooga Group, Inc.) with inactive probe will be used to deliver sham massage.
  Arms: Control Group
Procedure: Medium-Intensity Roller Massage — This group will receive a single bout of roller massage at medium intensity (25 newtons of force directed perpendicular to the surface of the thigh).
  Arms: Medium-Intensity Roller Massage
Procedure: High-Intensity Roller Massage — This group will receive a single bout of roller massage at medium intensity (45 newtons of force directed perpendicular to the surface of the thigh).
  Arms: High-Intensity Roller Massage

SUMMARY:
Muscle stiffness is associated with a variety of variables that affect health, however there is limited research on the effect of massage on muscle stiffness, and existing research does not quantify the intensity of massage. Thus trial will determine the effect of roller massage on quadriceps muscle stiffness and passive range of motion.

DETAILED DESCRIPTION:
Following screening for eligibility and consent, subjects will be assigned randomly to one of three groups: a placebo control group and two roller massage groups (treatment groups). The treatment groups will each receive a single bout of roller massage. One treatment group will receive a massage at medium intensity (25 newtons of force directed perpendicular to surface of thigh), the other treatment group at high intensity (45 newtons of force directed perpendicular to surface of thigh). The placebo group will receive a single bout of sham ultrasound. Both placebo and treatments will be delivered to the anterior thigh with the participant in a supine position. Each procedure will last for 10 minutes. In all groups, muscle stiffness, natural oscillation frequency, elasticity, relaxation time, and creep at the vastus lateralis will be measured using a myotonometer. PROM for knee flexion will also be measured in both groups using goniometry. All measurements will be taken at 3 different times: immediately before treatment or placebo, immediately after treatment or placebo, and 30 minutes after treatment or placebo. Myotonometric measurements of the vastus lateralis will be taken 2/3 of the way down between the anterior superior iliac spine and lateral aspect of the patella, in accordance with guidelines for the Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles. For goniometric measurement, participants will be in supine position on an examination table. The investigator will flex the participant's hip to 90 degrees and then, using a dynamometer (to ensure consistent applied force for all participants), flex the participant's knee. To measure knee flexion PROM, the goniometer will be positioned with the axis at the lateral epicondyle of the femur, the stationary arm in line with the lateral midline of the femur toward the greater trochanter, and the moving arm in line with the fibular head and lateral malleolus. During the time between the second and third measurements, subjects will be asked to sit quietly.

ELIGIBILITY:
Inclusion Criteria:

-Age 18-30

Exclusion Criteria:

* Prior history of significant vascular or neuromuscular illness or impairment affecting the lower limbs
* Serious injuries to the back or legs in the last six months
* Discomfort or pain in the back or legs
* Use of pain and anti-inflammatory medications
* Any contraindications to massage treatment or ultrasound
* Body mass index (BMI) >30 kg/m2.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Change in Quadriceps Stiffness | 1 hour (at baseline, immediately after treatment and 30 minutes later)
  Quadriceps stiffness will be measured using a myotonometer at baseline, immediately after treatment, and 30 minutes later.
Change in Passive Range of Motion | 1 hour (at baseline, immediately after treatment and 30 minutes later)
  Range of motion of the knee will be measured using a goniometer at baseline, immediately after treatment, and 30 minutes later.

SECONDARY OUTCOMES:
Change in Quadriceps Natural Oscillation Frequency | 1 hour (at baseline, immediately after treatment and 30 minutes later)
  Quadriceps natural oscillation frequency will be measured using a myotonometer at baseline, immediately after treatment, and 30 minutes later.
Change in Quadriceps Elasticity | 1 hour (at baseline, immediately after treatment and 30 minutes later)
  Quadriceps elasticity will be measured using a myotonometer at baseline, immediately after treatment, and 30 minutes later.
Change in Quadriceps Relaxation Time | 1 hour (at baseline, immediately after treatment and 30 minutes later)
  Quadriceps relaxation time will be measured using a myotonometer at baseline, immediately after treatment, and 30 minutes later.
Change in Quadriceps Creep | 1 hour (at baseline, immediately after treatment and 30 minutes later)
  Quadriceps creep will be measured using a myotonometer at baseline, immediately after treatment, and 30 minutes later.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Sykora, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No